CLINICAL TRIAL: NCT06131333
Title: Complex Coronary Artery Disease Treated With Percutaneous Coronary Intervention - COMPLEX Registry.
Brief Title: Complex CAD Treated With PCI With DES Implantation.
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sylwia Iwanczyk, Principal Investigator, Poznan University of Medical Sciences
Other Study IDs: 821/23
Record Dates: First submitted 2023-10-26; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Complex Coronary Artery Disease
MeSH Terms: interventions — Percutaneous Coronary Intervention; Drug Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complex PCI: All consecutive patients with complex coronary artery disease (CAD) were treated with percutaneous coronary intervention (PCI). The complexity of CAD was defined as having at least one of the following characteristics: chronic total occlusion (CTO), lesion length >40 mm, severe calcification assessed by angiography or intravascular imaging examination, multivessel PCI during the same intervention, or true bifurcation defined as any lesion involving both the main vessel (MV), proximal or distal and the ostium of the side branch (SB) (Medina 1,1,1; 1,0,1; or 0,1,1).
  Interventions: Procedure: Percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation — PCI was performed according to the general and local recommendations. The choice of DES among the new generation DES and the decision on procedure optimization belonged to the operator.

SUMMARY:
COMPLEX Registry is an investigator-initiated, retrospective, high-volume Polish single-center clinical registry enrolling 980 consecutive patients with complex coronary artery lesions treated percutaneously between September 2015 and December 2021. All data were collected prospectively as regards the clinical and technical endpoints. The study aimed to assess the safety and efficacy of new-generation, thin-struts DES in patients with complex CAD at long-term clinical follow-up. The primary endpoint of the study was the occurrence of TLR during follow-up. Secondary endpoints were a procedural success and the occurrence of MACE, including all-cause death, MI, or TLR.

ELIGIBILITY:
Inclusion Criteria:

* For the inclusion of patients in this study, the complexity of CAD was defined as having at least one of the following characteristics: chronic total occlusion (CTO), lesion length >40 mm, severe calcification assessed by angiography or intravascular imaging examination, multivessel PCI during the same intervention, or true bifurcation defined as any lesion involving both the main vessel (MV), proximal or distal and the ostium of the side branch (SB) (Medina 1,1,1; 1,0,1; or 0,1,1).

Exclusion Criteria:

* left main stem
* PCI treated during index procedure;
* cardiogenic shock,
* thrombolysis before PCI;
* 12-month follow-up not available

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with symptomatic CAD, including chronic coronary syndromes (CCS) and acute coronary syndromes (ACS), qualified for PCI and meeting the criteria for complex CAD were included in the analysis.
Sampling Method: Probability Sample
Enrollment: 980 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Target lesion revascularization (TLR) | 12 months
  During the 12-month follow-up, the incidence of TLR in patients included in the study will be reported. TLR was defined as revascularization post-stenting within the stent or within the 5-mm borders adjacent to the stent.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 12 month
  During the 12-month follow-up, the incidence of MACE in patients included in the study will be assessed. Major adverse cardiac event composed of all-cause death, myocardial infarction (MI), or TLR.
Procedural success | Peri-procedural
  Procedural success was defined as angiographic success in the absence of in-hospital major events including death, MI, need for TLR, stroke, vascular access site complications, and contrast agent nephropathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Medical Sciences, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided